CLINICAL TRIAL: NCT06106165
Title: Improving Uptake of Breast, Bowel and Cervical Cancer Screening Among Muslim Women: a Non-randomised Feasibility Study of a Peer-led, Faith-based Intervention
Brief Title: Improving Muslim Women's Uptake of Cancer Screening (IMCAN)
Acronym: IMCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sunderland (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Floor Christie-de Jong, Senior lecturer, University of Sunderland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EDDPJT-May22\100030
Record Dates: First submitted 2023-08-16; First posted 2023-10-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Bowel Cancer; Cervical Cancer
Keywords: Cancer screening; Breast Cancer; Bowel Cancer; Cervical Cancer; Faith-based intervention; Muslim women
MeSH Terms: conditions — Breast Neoplasms; Intestinal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-person delivery (Experimental): Participants will attend the workshops in a mosque or community centre.
  Interventions: Other: In-person peer-led faith-based intervention to encourage breast, bowel, and cervical screening uptake among Muslim women
- Online delivery (Experimental): Participants will join the workshops via a web conferencing platform The content of the online workshops is identical to the content of in-person workshops.
  Interventions: Other: Online In-person peer-led faith-based intervention to encourage breast, bowel, and cervical screening uptake among Muslim women

INTERVENTIONS:
Other: In-person peer-led faith-based intervention to encourage breast, bowel, and cervical screening uptake among Muslim women — The intervention includes a two-hour workshop, delivered in-person, that aims to improve the uptake of cancer screening among Muslim women.
  The workshop consists of four parts:
  * A peer-led discussion on barriers and facilitators to breast, cervical and colorectal cancer screening
  * A health information session led by a health professional
  * Videos of Muslim women talking about their experiences with cancer screening
  * A religious perspective on cancer screening led by a female religious scholar
  Arms: In-person delivery
Other: Online In-person peer-led faith-based intervention to encourage breast, bowel, and cervical screening uptake among Muslim women — The intervention includes a two-hour workshop, delivered online, that aims to improve the uptake of cancer screening among Muslim women.
  The workshop consists of four parts:
  * A peer-led discussion on barriers and facilitators to breast, cervical and colorectal cancer screening
  * A health information session led by a health professional
  * Videos of Muslim women talking about their experiences with cancer screening
  * A religious perspective on cancer screening led by a female religious scholar
  Arms: Online delivery

SUMMARY:
The goal of this non-randomised trial is to test how a workshop that includes religiously-tailored messages can help increase the uptake of breast, colorectal and cervical cancer screening among Muslim women in North East England and Scotland.

The results of this trial will inform the development of a full-scale randomised-controlled trial.

Participants in this study will be asked to take part in a two-hour workshop, deliver either online or in-person.

DETAILED DESCRIPTION:
Low rates of cancer screening among Muslim women puts them at higher risk of death from screening since they do not detect cancer early. This study will work to increase the uptake of cancer screening among Muslim women using two-hour workshops delivered in the community.

The workshops were developed with the help of 10 Muslim women in Scotland. The workshops include four parts:

* A discussion on the barriers and facilitators to breast, cervical and colorectal cancer screening
* A health information session given by a female health provider on cancer screening
* Videos of Muslim women talking about their experiences with cancer screening
* A session given by a female religious scholar to discuss Islamic perspectives on cancer screening.

Another eighteen Muslim women then took part in the workshops; they gave positive feedback on the content of the workshops and how the sessions were delivered.

In the feasibility trial, the workshops will be delivered to 200 Muslim women to find out whether a full-scale randomised-controlled trial can take place. This study will be carried out with the help of 10 Muslim women who will give advice on the content of the workshops and plan for implementation; they will also help with the delivery of the workshops.

It is expected that this study will lead to changes in knowledge and screening uptake among participants.

ELIGIBILITY:
Inclusion Criteria:

* Women from any ethnicity identifying as Muslim
* Muslim Women aged 25-74 years
* Muslim women living in North East England or Scotland
* Muslim women who are not up-to-date with all cancer screening they are eligible for; women who are up-to-date with one type of screening but not others would be eligible (for example, women might be up-to-date with breast cancer screening but not cervical or bowel cancer screening)

Exclusion Criteria:

* Women who do not identify as Muslim
* Women aged less than 25 years or older than 74 years
* Women who are up-to-date with all the screening they are eligible for
* Women who had either breast, cervical or bowel cancer before as their knowledge of the disease and treatment would differ from other women who do not have any prior experience with the disease
* Women who have had BReast CAncer gene testing and underwent mastectomy and/or hysterectomy

Ages: 25 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Narrative description of feasibility | 12 months
  The primary outcome of the project will be a narrative description of study feasibility, including recruitment and retention, protocol adherence and stakeholder acceptability. The primary outcome will be assessed using a mixed methods approach and assessed according the progression criteria, as described below.
Recruitment feasibility | Baseline, 5 months, 7 months, 12 months
  Determine how many women accept the invitation to participate in the study and to estimate eligibility, recruitment and refusal rates.
  This will be assessed using project monitoring data maintained by the research team which logs in detail all study data, including number of people, time, missing data, and cost where relevant.
  Eligibility rate: Calculated as the number of participants screened/number of participants eligible x100%
  Recruitment rate: Calculated as the number of enrolled participants/number of eligible participants x 100%
  We will report recruitment and retention rates with 90% confidence intervals. Recruitment and retention rates will be summarised in relation to baseline characteristics, and differences in retention rates will be assessed using logistic regression methods.
Screening status of participants and the proportion of participants who were partially/not up to date with screening | Baseline
  Estimate the screening-non-responder rate. Non-responder rate: Calculated as the number of enrolled participants who were screening non-responders/number of eligible participants x 100%
Retention rate | 6 months, 12 months
  Estimate loss to follow up/retention rate.
  This will be assessed using project monitoring data Retention rate: Calculated as the number of participants who complete the 12 months follow up/number of participants in the intervention x100% This data will be compared for non-responders and partial responders.
Peer educator recruitment feasibility | baseline, 12 months
  Number of women who accepted the invitation to become peer educators, and the number of peer educators retained at 12 months. This will be assessed using project monitoring data.
  Peer-educator recruitment rate: Calculated as the number of enrolled peer-educators/number of eligible peer-educators x 100% Peer-educator retention rate: calculated as the number of peer-educators at 12 months/number of peer-educators recruited x 100%
Feasibility of obtaining screening data | 12 months
  Whether the research team was able to obtain screening records for participants in all study location, and the proportion of participants who gave consent to access their screening records
Questionnaire response rate | Baseline, 6 months, 12 months
  The proportion of participants responding to questionnaires at baseline, 6 months and 12 months.
Feasibility of measuring secondary outcomes | Baseline, 6 months, 12 months
  Measure key secondary outcome measures including behavioural intention proxies, and feasibility of self-reported data, missing data, estimates, variances and 95% CIs for any comparisons.
  Baseline and follow up data
  Data will be assessed in relation to each of the 3 different types of screening, as well as generally, to ensure we capture whether the intervention has a differential impact on different screening types.
  We will also aim to compare behavioural change and self-reported data with the actual NHS screening data.
  Participants' scores on outcome scales, and changes over time, will be reported using descriptive methods. Paired t-tests, or non-parametric alternatives, will be used to estimate changes over time, with 90% confidence intervals. Correlations between baseline and follow-up measures will be reported with 90% confidence intervals.
Difference on key domains between intervention modalities (online/face to face) | Baseline, 6 months, 12 months
  Comparison of measures on key domains for trial parameters will provide insight into the feasibility of the two different modes of delivery.
  This will be inspected using project monitoring data baseline and follow up measures.
  Including: eligibility rate, recruitment rate, retention rate, all measures non-responders/attenders and missing data
  Visual inspection of trends and descriptive data will be used to establish whether comparisons between modalities is feasible.
The acceptability of the study engagement process to peer-educators | 12 months
  Qualitative exploration of the acceptability of the process of recruitment, co-design phase, training, experiences and delivery of intervention.
  Qualitative process evaluation focus groups with peer-educators. Including: experiences of co-design phase, experiences of recruitment of peer-educators, experiences of training, experiences of delivery of the intervention, language and use of interpreters, and perspectives on the intervention and study.
The acceptability of the intervention and its implementation to participants and stakeholders, including intervention components and delivery mode (online/face-to-face) | 12 months
  Qualitative exploration of the acceptability of the intervention and its delivery with participants and key stakeholders.
  Qualitative process evaluation focus groups with participants and interviews with stakeholders.
  This explores the following: content of the intervention, delivery mode of the intervention (face-to-face/online), delivery of the intervention (peer-educators, health care provider, religious perspective, personal testimonials), and experience and perspectives of taking part in the intervention
The acceptability of data collection methods used to participants and stakeholders | 12 months
  Qualitative exploration of the acceptability of the data collection methods and secondary outcome measures with participants and key stakeholders.
  Qualitative process evaluation focus groups with participants and interviews with stakeholders Including: invitation to participate , recruitment processes, consent taking, baseline and follow-up secondary outcome measures, engagement in baseline and follow-up processes, and willingness to be randomised.
Adherence to protocol | 12 months
  Explore qualitatively protocol adherence and barriers and enablers to key stakeholders such as research staff and collaborators. Qualitative process evaluation interviews with research staff and collaborators.

SECONDARY OUTCOMES:
Religious health fatalism questionnaire (RHFQ) | Baseline
  A questionnaire will be given to participants to test how religious beliefs influence health beliefs and willingness to obtain screening and medical treatments.
  RHFQ includes 8 statements that are answered on 5-point Likert scale: 1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree Higher scores indicate higher levels of religious fatalism, thus a lower willingness to attend screening due to religious beliefs
Modesty | Baseline
  The Modesty Measure for Muslim women (MMM-W) will be given to participants to examine how self-representation among Muslim women can affect their health seeking behaviours.
  The questionnaire will ask participants to indicate whether they 'agree', 'disagree' or 'ambivalent' to 10 statements about modest behaviour and healthcare
Sociodemographic descriptors | Baseline
  Participant characteristics, such as age, location, education level, ethnicity, professional occupation and marital status, will be recorded
Cancer knowledge questions adapted from Cancer Awareness Measures (CAM) by Cancer Research UK | baseline, 6 months and 12 months
  This measure will assess changes in knowledge about the risk factors, symptoms and screening of breast, bowel and cervical cancer among participants.
  The questionnaire will be administered online through Qualtrics (a telephone option will also be offered).
  Multiple choice questions are used for this measure.
Cancer screening behaviour | baseline, 6 months and 12 months
  A cancer screening behaviour questionnaire will be given to participants. This consists of 2 parts:
  1. Participants will be asked about whether they attended breast, bowel or cervical cancer screening and if they are planning to attend screening. The answers for these questions will be: 'yes', 'no' or 'I don't know'.
  2. The second part includes statements that represent barrier and facilitator beliefs that might affect screening behaviour. Participants will be asked to indicate the level of agreement with each statement on 5-point liker scale: 1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree
Self-reported screening uptake | baseline, 6 months and 12 months
  Change in the number of participants who obtained screening following the intervention. This outcome is self-reported by participants
Actual screening uptake | baseline, 6 months and 12 months
  Screening data from the National Health Services (NHS) will be analysed to examine the change in the number of participants who obtained screening following the intervention.
Quality of life measures | Baseline, 6 months, 12 months
  Intervention participants will be asked to fill EQ-5D-5L questionnaires, which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University of Glasgow, Glasgow, Scotland
  - University of Sunderland, Sunderland, Tyne and Wear